CLINICAL TRIAL: NCT05865795
Title: Mapping the Natural History of Parenychymal and Cerebral Perfusion Changes in Acute Ischemic and Hemorrhagic Strokes Using Cranial Ultrasound and Continuous Trans-Cranial Doppler
Brief Title: Mapping the Natural History of Parenychymal and Cerebral Perfusion Changes in Acute Ischemic and Hemorrhagic Strokes
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00048743
Record Dates: First submitted 2023-05-09; First posted 2023-05-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke; Hemorrhagic Stroke
Keywords: hypertension; hypotension; stroke therapy; cerebral perfusion
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Hypertension; Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study using ultrasound of the brain as a diagnostic tool to differentiate between ischemic stroke and hemorrhagic stroke. Correlation of brain perfusion and size of stroke in relation to systemic hemodynamic targets will be assessed on serial scans.

DETAILED DESCRIPTION:
To explore the correlation of brain parenchyma lesions changes and cerebral perfusion parameters as measured by cranial ultrasound transcranial Doppler to patient's blood pressure in a continuous fashion and correlate these to clinical and radiological features of cerebral perfusion. This study will lead to answering clinical management questions like is accurate diagnosis of hemorrhagic stroke possible that could be applied to the field evaluation of stroke patients, optimum blood pressure targets for different subsets of population studied ( multifocal disease, collateralized circulation etc), course of fluctuations in cerebral blood flow in response to systemic blood pressure changes or presence of persistent embolic signals in patients with presumed cardio-embolic strokes.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over the age of 18 who present to Wake Forest Baptist Hospital, get evaluated in the Emergency Department and /or admitted to inpatient/Intensive Care Unit and received any neuroimaging ordered by clinical team (head) (CT) (computerized tomography or Magnetic Resonance Imaging) (MRI) with diagnosis of acute ischemic or hemorrhagic strokes or stroke mimic or suspicion of intracranial pathology

Exclusion Criteria:

* Patients with Age < 18
* Incarcerate and Pregnant patients
* Penetrating cranial/head trauma or scalp wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting with stroke like presentation and suspicion of intracranial pathology will be screened on presentation to the Emergency Department and/or admission to WFBMC. Many pathologies look like strokes on presentation hence included as controls. Exclusion criteria will be age < 18, pregnant, incarcerated patients, or any scalp/cranial/ penetrating head trauma.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Collection of Images | Baseline
  To explore the systemic hemodynamic correlates of cerebral blood flow parameters following acute ischemic and/or hemorrhagic strokes in relation to lesion size seen in B mode images.

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Sarwal, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee